CLINICAL TRIAL: NCT01174030
Title: A 4-week, Randomized, Double-blind, Parallel-group, Vehicle-controlled, Multicenter Study Investigating the Efficacy and Safety of CD07805/47 Gel 0.5% Applied Topically Once Daily (QD), and CD07805/47 Gel 0.18% Applied Topically Once Daily (QD) or Twice Daily (BID), in Subjects With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: Efficacy and Safety Study of CD07805/47 Topical Gel in Subjects With Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.18161
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2014-01

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- CD07805/47 Gel 0.5% QD (Experimental)
  Interventions: Drug: CD07805/47 Gel
- CD07805/47 Gel 0.18% QD (Experimental)
  Interventions: Drug: CD07805/47 Gel
- CD07805/47 Gel 0.18% BID (Experimental)
  Interventions: Drug: CD07805/47 Gel
- Vehicle Gel QD (Placebo Comparator)
  Interventions: Drug: Vehicle Gel
- Vehicle Gel BID (Placebo Comparator)
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: CD07805/47 Gel — CD07805/47 Gel 0.5% QD
  Arms: CD07805/47 Gel 0.5% QD
Drug: Vehicle Gel — Vehicle Gel QD
  Arms: Vehicle Gel QD
Drug: CD07805/47 Gel — CD07805/47 Gel 0.18% QD
  Arms: CD07805/47 Gel 0.18% QD
Drug: CD07805/47 Gel — CD07805/47 Gel 0.18% BID
  Arms: CD07805/47 Gel 0.18% BID
Drug: Vehicle Gel — Vehicle Gel BID
  Arms: Vehicle Gel BID

SUMMARY:
The purpose of this vehicle controlled study is to evaluate the efficacy and safety of CD07805/47 gel 0.5% applied topically once daily (QD) for 4 weeks, and CD07805/47 gel 0.18% applied topically once daily (QD) or twice daily (BID) for 4 weeks, in subjects with moderate to severe facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, who is at least 18 years of age or older.
* A clinical diagnosis of rosacea.
* A Clinician Erythema Assessment (CEA) score of 3 at Screening and at Pre-dose (T0) on Baseline/Day 1.
* A Patient Self Assessment-5 (PSA-5) score of 3 at Screening and at Pre-dose (T0) on Baseline/Day 1.
* A Patient Self Assessment-11 (PSA-11) score of 5 at Screening and at Pre-dose (T0) on Baseline/Day 1.

Exclusion Criteria:

* Three (3) or more facial inflammatory lesions.
* Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression.
* Known allergies or sensitivities to any components of the study medications, including the active gel ingredient, brimonidine tartrate.
* Intraocular pressure (IOP) measurement less than 10 mm Hg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D, Inc; William Abramovits, MD, Principal Investigator — Dermatology Treatment & Research Center; Fran Cook-Bolden, MD, Principal Investigator — Skin Specialty Group; Zoe Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, PSC; Kimberly Grande, MD, Principal Investigator — The Skin Wellness Center; Michael Heffernan, MD, Principal Investigator — Central Dermatology PC; Steven Kempers, MD, Principal Investigator — Minnesota Clinical Study Center; Mark Ling, MD, Principal Investigator — Meda Phase, Inc.; Robert Matheson, MD, Principal Investigator — Oregon Medical Research; Kappa Meadows, MD, Principal Investigator — The Education & Research Foundation; Angela Moore, MD, Principal Investigator — Arlington Center for Dermatology; Girish Munavalli, MD, Principal Investigator — Dermatology, Laser & Vein Specialists of the Carolinas; Andrew Pollack, MD, Principal Investigator — Philadelphia Institute of Dermatology; Phoebe Rich, MD, Principal Investigator — Oregon Dermatology & Research Center; Harry Sharta, MD, Principal Investigator — Madison Skin & Research; Martin Steinhoff, MD, Principal Investigator — University of California at San Francisco; Dow Stough, MD, Principal Investigator — Burke Pharmaceutical Research; William Werschler, MD, Principal Investigator — Premier Clinical Research; Patricia Westmoreland, MD, Principal Investigator — Palmetto Clinical Trial Services, LLC; Stephen Schleicher, MD, Principal Investigator — DermDox
Locations (20):
- United States (20):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - University of California at San Francisco, San Francisco, California
  - Meda Phase, Inc, Newnan, Georgia
  - Dermatology Specialists PC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Central Dermatology, PC, St Louis, Missouri
  - Skin Specialty Group, New York, New York
  - Dermatology Laser & Vein Specialists, Charlotte, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Oregon Medical Research, Portland, Oregon
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - DermDox, Hazleton, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - The Skin Wellness Center, Knoxville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Dermatology Treatment & Research Center, Dallas, Texas
  - The Education & Research Foundation, Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington
  - Madison Skin & Research, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- CD07805/47 Gel 0.5% QD: CD07805/47 Gel 0.5% Once Daily
- CD07805/47 Gel 0.18% QD: CD07805/47 Gel 0.18% Once Daily
- CD07805/47 Gel 0.18% BID: CD07805/47 Gel 0.18% Twice Daily
- Vehicle Gel QD: Vehicle Gel Once Daily
- Vehicle Gel BID: Vehicle Gel Twice Daily
Period: Overall Study
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID
Started | 53 | 54 | 54 | 55 | 53
Completed | 51 | 52 | 52 | 53 | 52
Not Completed | 2 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID | Total
Number analyzed (Participants) | 53 | 54 | 54 | 55 | 53 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 50 | 50 | 54 | 51 | 257
  >=65 years | 1 | 4 | 4 | 1 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.50) | 46.9 (12.72) | 43.2 (12.28) | 43.4 (12.73) | 43.0 (12.33) | 44.3 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 42 | 45 | 44 | 217
  Male | 11 | 10 | 12 | 10 | 9 | 52
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 54 | 55 | 53 | 269

OUTCOME MEASURES:

1. Primary Outcome: Composite Success
Description: Composite success defined as 2-grade improvement on Clinician Erythema Assessment (CEA)and Patient Self Assessment-5 (PSA-5).
  Each concentration/regimen was compared to its respective placebo control as part of the primary analysis.
Time Frame: Day 29
Population: Intent-to Treat (ITT) population, LOCF when the data are missing at all four timepoints (i.e. Hours 3, 6, 9, 12) LOCF method will be applied from previous visit.
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID
Number analyzed (Participants) | 53 | 54 | 54 | 55 | 53
participants
  Day 29/Hour 3 | 16 | 10 | 10 | 2 | 4
  Day 29/Hour 6 | 15 | 10 | 9 | 4 | 7
  Day 29/Hour 9 | 17 | 7 | 11 | 2 | 10
  Day 29/Hour 12 | 10 | 5 | 8 | 2 | 9
Statistical Analysis 1: Comparison: CD07805/47 Gel 0.5% QD vs Vehicle Gel QD; Test type: Superiority or Other; p < 0.001, GEE:Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 8.392, 95% CI [2.637 to 26.710]
Statistical Analysis 2: Comparison: CD07805/47 Gel 0.18% BID vs Vehicle Gel BID; Test type: Superiority or Other; p = 0.549, GEE:Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 1.269, 95% CI [0.586 to 2.747]
Statistical Analysis 3: Comparison: CD07805/47 Gel 0.18% QD vs Vehicle Gel QD; Test type: Superiority or Other; p = 0.027, GEE:Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 3.738, 95% CI [1.097 to 12.742]

2. Secondary Outcome: CEA Success
Description: CEA success defined as 2-grade improvement on CEA.
  Each concentration/regimen was compared to its respective placebo control as part of the primary analysis.
  Clinician Erythema Assessment (CEA) - Grade/Description 0 / Clear Skin with no signs of erythema
  1. / Amost clear; slight redness
  2. / Mild erythema; definite redness
  3. / Moderate erythema; marked redness
  4. / Severe erythema; fiery redness
Time Frame: Day 29
Population: ITT population, LOCF when the data are missing at all four timepoints (i.e. Hours 3,6,9,12) LOCF method will be applied from the previous visit.
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID
Number analyzed (Participants) | 53 | 54 | 54 | 55 | 53
participants
  Day 29/Hour 3 | 27 | 21 | 22 | 12 | 9
  Day 29/Hour 6 | 23 | 21 | 18 | 12 | 12
  Day 29/Hour 9 | 26 | 20 | 23 | 12 | 15
  Day 29/Hour 12 | 20 | 17 | 18 | 12 | 16
Statistical Analysis 1: Comparison: CD07805/47 Gel 0.5% QD vs Vehicle Gel QD; Test type: Superiority or Other; p = .003, GEE:Logit link Function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 2.683, 95% CI [1.388 to 5.188]
Statistical Analysis 2: Comparison: CD07805/47 Gel 0.18% BID vs Vehicle Gel BID; Test type: Superiority or Other; p = 0.056, GEE: Logit link Function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 1.892, 95% CI [0.980 to 3.651]
Statistical Analysis 3: Comparison: CD07805/47 Gel 0.18% QD vs Vehicle Gel QD; Test type: Superiority or Other; p = 0.074, GEE:Logit link Function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 1.885, 95% CI [0.946 to 3.756]

3. Secondary Outcome: PSA-5 Success
Description: Each concentration/regimen was compared to its respective placebo control as part of the primary analysis.
  PSA-5 success defined as 2-grade improvement on PSA-5.
  Patient Self Assessment - 5 (PSA-5) - Grade/description 0 / No redness
  1. / Very mild redness
  2. / Mild redness
  3. / Moderate redness
  4. / Severe redness
Time Frame: day 29
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID
Number analyzed (Participants) | 53 | 54 | 54 | 55 | 53
participants
  Day 29/Hour 3 | 25 | 17 | 20 | 7 | 11
  Day 29/Hour 6 | 26 | 13 | 15 | 8 | 11
  Day 29/Hour 9 | 22 | 9 | 19 | 5 | 13
  Day 29/Hour 12 | 20 | 9 | 16 | 5 | 10
Statistical Analysis 1: Comparison: CD07805/47 Gel 0.5% QD vs Vehicle Gel QD; Test type: Superiority or Other; p < 0.001, GEE: Logit link function; Generalize Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 6.582, 95% CI [2.755 to 15.723]
Statistical Analysis 2: Comparison: CD07805/47 Gel 0.18% BID vs Vehicle Gel BID; Test type: Superiority or Other; p = 0.093, GEE: Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 1.853, 95% CI [0.903 to 3.802]
Statistical Analysis 3: Comparison: CD07805/47 Gel 0.18% QD vs Vehicle Gel QD; Test type: Superiority or Other; p = 0.054, GEE: Logit link function; Generalized Estimating Equation (GEE) methods with Logit link function and marginal expectation model; Odds Ratio (OR) = 2.365, 95% CI [0.960 to 5.825]

ADVERSE EVENTS:
Arm/Group | CD07805/47 Gel 0.5% QD | CD07805/47 Gel 0.18% QD | CD07805/47 Gel 0.18% BID | Vehicle Gel QD | Vehicle Gel BID
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/54 | 0/54 | 1/55 | 0/53
Other Adverse Events (participants affected / at risk) | 18/53 | 13/54 | 14/54 | 16/55 | 8/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 Gel 0.5% QD (N=53) | CD07805/47 Gel 0.18% QD (N=54) | CD07805/47 Gel 0.18% BID (N=54) | Vehicle Gel QD (N=55) | Vehicle Gel BID (N=53)
Gastric Reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 Gel 0.5% QD (N=53) | CD07805/47 Gel 0.18% QD (N=54) | CD07805/47 Gel 0.18% BID (N=54) | Vehicle Gel QD (N=55) | Vehicle Gel BID (N=53)
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 4 | 0
Flushing (Vascular disorders) | 4 | 1 | 0 | 0 | 0
Intraocular pressure increased (Eye disorders) | 7 | 6 | 8 | 9 | 4
Headache (Nervous system disorders) | 4 | 3 | 3 | 1 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 1 | 0
Skin Warm (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days